CLINICAL TRIAL: NCT05934292
Title: An Open-Label, Single-Dose Clinical Study to Evaluate the Pharmacokinetics of MK-0616 in Participants With Varying Degrees of Renal Impairment
Brief Title: Enlicitide Decanoate (MK-0616 Oral PCSK9 Inhibitor) Renal Impairment Study (MK-0616-020)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0616-020; MK-0616-020 (Other: MSD)
Record Dates: First submitted 2023-06-05; First posted 2023-07-06 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Panel A: Moderate Renal Impairment (RI) (Experimental): Participants receive Enlicitide Decanoate 20 mg tablet single dose orally on Day 1
  Interventions: Drug: Enlicitide Decanoate
- Panel B: Severe RI (Experimental): Participants receive Enlicitide Decanoate 20 mg tablet single dose orally on Day 1
  Interventions: Drug: Enlicitide Decanoate
- Panel C: End-Stage Renal Disease (ESRD) on Hemodialysis (HD) (Experimental): Participants receive Enlicitide Decanoate 20 mg tablet orally on Day 1 and Day 16.
  Interventions: Drug: Enlicitide Decanoate
- Panel D: Healthy Controls (Experimental): Participants receive Enlicitide Decanoate 20 mg tablet single dose orally on Day 1.
  Interventions: Drug: Enlicitide Decanoate

INTERVENTIONS:
Drug: Enlicitide Decanoate — Oral dose
  Other Names: MK-0616

SUMMARY:
The primary objective of the study is to compare the plasma pharmacokinetics (PK) of enlicitide decanoate following a single 20 mg dose in participants on a background of statin therapy with varying degrees of renal impairment (moderate, severe, end stage renal disease [ESRD]) to those of healthy mean matched control participants on a background of statin therapy. There is no formal hypothesis.

DETAILED DESCRIPTION:
Panel C included participants with ESRD. No urine samples could be obtained on Panel C participants and hence no pharmacokinetic (PK) analysis could be performed for Panel C participants as pre-specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Be in good health with the exception of renal impairment (RI) and hypercholesterolemia for participants in Panels A, B, and C. Participants with RI that have stable, chronic medical or psychiatric conditions, including but not limited to hypertension, hypercholesterolemia, diabetes mellitus, hyper- or hypothyroidism, gout, and chronic anxiety or depression may be included at the discretion of the investigator
* Body Mass Index (BMI) ≥ 18 kg/m^2 and ≤ 40 kg/m^2, inclusive
* Be on a stable dose of any statin therapy defined as: no changes to dose or type of statin therapy for at least 2 months prior to Screening and participant anticipates no changes to statin therapy throughout the study until the poststudy visit

Exclusion Criteria:

* History or presence of renal artery stenosis
* Had a functioning renal transplant in the past 5 years and is taking transplant medication
* Participants in panels A, B and D: Has rapidly fluctuating renal function as determined by historical measurements
* Has a history gastrointestinal disease which might affect food and drug absorption, as determined by the investigator, or has had gastric bypass or similar surgery
* History of cancer (malignancy)
* History of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food
* Has received an anti-proprotein convertase subtilisin/kexin type 9 (PCSK9) small molecule treatment, monoclonal antibody, or short interfering RNA (siRNA) or RNA interference (ie, Inclisiran) within 12 months prior to Screening
* Participants with RI (Panels A, B, and C): Taking medications to treat chronic medical conditions and/or conditions associated with renal disease, if participant has not been on a stable regimen for at least 1 month (other than statins, which require a stable dose for at least 2 months) prior to administration of the initial dose of study intervention, and/or is unable to withhold the use of the medication(s) within 4 hours prior to and 4 hours after administration of study intervention
* Participated in another investigational study within 4 weeks prior to the prestudy (screening) visit
* Consumes greater than 3 servings of alcoholic beverages per day
* Consumes excessive amounts, defined as greater than 6 servings of caffeinated beverages per day

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- United States (5):
  - Velocity Clinical Research, Hallandale Beach ( Site 0003), Hallandale, Florida
  - Clinical Pharmacology of Miami ( Site 0005), Miami, Florida
  - Advanced Pharma CR, LLC ( Site 0001), Miami, Florida
  - Orlando Clinical Research Center ( Site 0004), Orlando, Florida
  - Genesis Clinical Research, LLC ( Site 0002), Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All allocated participants. Panel C included participants with End-Stage Renal Disease (ESRD). No urine samples could be obtained on Panel C participants and hence no pharmacokinetic (PK) analysis could be performed for Panel C participants as pre-specified in the protocol.
Groups:
- Panel A: Moderate Renal Impairment (RI); Panel B: Severe RI; Panel D: Healthy Controls: Participants received Enlicitide Decanoate 20 mg tablet single dose orally on Day 1.
- Panel C: End-Stage Renal Disease (ESRD) on Hemodialysis (HD): Participants received Enlicitide Decanoate 20 mg tablet orally on Day 1 and Day 16.
Period: Overall Study
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: End-Stage Renal Disease (ESRD) on Hemodialysis (HD) | Panel D: Healthy Controls
Started | 8 | 8 | 9 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All allocated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: End-Stage Renal Disease (ESRD) on Hemodialysis (HD) | Panel D: Healthy Controls | Total
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67 (9.6) | 66.8 (12.1) | 60.1 (9.6) | 62.8 (4) | 64 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 2 | 9
  Male | 7 | 3 | 8 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 2 | 5 | 15
  Not Hispanic or Latino | 2 | 6 | 7 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 7 | 3 | 16
  White | 7 | 3 | 2 | 5 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-Inf) of Enlicitide Decanoate
Description: AUC0-inf was a measure of the total amount of drug in the plasma from the dose administration extrapolated to infinity. Blood for plasma samples was collected at pre-specified timepoints to determine the AUC0-inf of enlicitide decanoate for Panel A, B, C, and D participants. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C ESRD - enlicitide decanoate pre-hemodialysis and Panel C ESRD - enlicitide decanoate post-hemodialysis to report AUC0-inf. Per protocol, mean AUC0-inf was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 120, 168, and 240 hours postdose
Population: All allocated participants of Panel A, B, C, and D who received at least a dose of study treatment and had data available for AUC0-inf.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*nmol/Liter
Groups:
- Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis: Participants received Enlicitide Decanoate 20 mg tablet orally on Day 1.
- Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis: Participants received Enlicitide Decanoate 20 mg tablet orally on Day 16.
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 8
hr*nmol/Liter | 733 [499 to 1080] | 554 [379 to 809] | 850 [538 to 1350] | 570 [404 to 804] | 487 [316 to 752]
Statistical Analysis 1: Comparison: Panel A: Moderate Renal Impairment (RI) vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 1.50, 90% CI 2-sided [0.98 to 2.31] — Geometric mean ratio (GMR) and 90% confidence interval (CI) were calculated using a linear fixed effects model performed on natural log-transformed values. GMR: Panel A-Moderate Renal Impairment (RI)/Panel D-Healthy controls
Statistical Analysis 2: Comparison: Panel B: Severe RI vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio; Geometric Mean Ratio = 1.14, 90% CI 2-sided [0.74 to 1.74] — GMR and 90% confidence interval (CI) were calculated using a linear fixed effects model performed on natural log-transformed values. GMR: Panel B-Severe RI/Panel D-Healthy controls
Statistical Analysis 3: Comparison: Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 1.75, 90% CI 2-sided [1.10 to 2.78] — GMR and 90% CI were calculated using a linear fixed effects model performed on natural log-transformed values. GMR: Panel C-ESRD Enlicitide Decanoate Pre-Hemodialysis/ Panel D-Healthy Controls
Statistical Analysis 4: Comparison: Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 1.17, 90% CI 2-sided [0.77 to 1.77] — GMR and 90% CI were calculated using a linear fixed effects model performed on natural log-transformed values. GMR: Panel C-ESRD Enlicitide Decanoate Post-Hemodialysis/ Panel D-Healthy Controls

2. Primary Outcome: AUC From Time 0 to Last Measurable Concentration (AUClast) of Enlicitide Decanoate
Description: AUClast was defined as the area under the concentration-time curve of enlicitide decanoate from time zero to last measurable concentration. Blood for plasma samples was collected at pre-specified timepoints to determine the AUClast of enlicitide decanoate in Panel A, B, C, and D participants. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C ESRD - enlicitide decanoate pre-hemodialysis and Panel C ESRD - enlicitide decanoate post-hemodialysis to report AUClast. Per protocol, mean AUClast was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 120, 168, and 240 hours postdose
Population: All participants of Panel A, B, C, and D who received at least a dose of study treatment and had data available for AUClast.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*nmol/Liter
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8
hr*nmol/Liter | 735 [506 to 1070] | 362 [145 to 904] | 649 [343 to 1230] | 538 [376 to 769] | 456 [297 to 701]
Statistical Analysis 1: Comparison: Panel A: Moderate Renal Impairment (RI) vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 1.61, 90% CI 2-sided [1.05 to 2.46] — GMR and 90% confidence interval (CI) were calculated using a linear fixed effects model performed on natural log-transformed values. GMR: Panel A-Moderate Renal Impairment (RI)/Panel D-Healthy controls
Statistical Analysis 2: Comparison: Panel B: Severe RI vs Panel D: Healthy Controls; Test type: Other; Geometric Mean ratio = 0.79, 90% CI 2-sided [0.37 to 1.72] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 1.42, 90% CI 2-sided [0.80 to 2.54] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 1.18, 90% CI 2-sided [0.78 to 1.78] — [estimate comment as in outcome 1, analysis 4]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Enlicitide Decanoate
Description: Cmax was defined as the maximum or peak concentration of enlicitide decanoate observed after its administration. Blood for plasma samples was collected at pre-specified time points to determine the Cmax of enlicitide decanoate in Panel A, B, C and D participants. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis to report Cmax. Per protocol, mean Cmax was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 120, 168, and 240 hours postdose
Population: All participants of Panel A, B, C, and D who received at least a dose of study treatment and had data available for Cmax.
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/Liter
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8
nmol/Liter | 9.56 [6.95 to 13.2] | 5.8 [3.03 to 11.1] | 8.73 [6.23 to 12.2] | 9.08 [6.13 to 13.4] | 9.72 [7.1 to 13.3]
Statistical Analysis 1: Comparison: Panel A: Moderate Renal Impairment (RI) vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.98, 90% CI 2-sided [0.71 to 1.37] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Panel B: Severe RI vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.60, 90% CI 2-sided [0.34 to 1.04] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.90, 90% CI 2-sided [0.64 to 1.27] — GMR and 90% confidence interval (CI) were calculated using a linear fixed effects model performed on natural log-transformed values. GMR: Panel C-ESRD Enlicitide Decanoate Pre-Hemodialysis/ Panel D-Healthy Controls
Statistical Analysis 4: Comparison: Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 1.18, 90% CI 2-sided [0.78 to 1.78] — GMR and 90% confidence interval (CI) were calculated using a linear fixed effects model performed on natural log-transformed values. GMR: Panel C-ESRD Enlicitide Decanoate Post-Hemodialysis/ Panel D-Healthy Controls

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Enlicitide Decanoate
Description: Tmax was defined as the time required for a study drug to reach maximum concentration in plasma. Blood for plasma samples was collected at pre-specified time points to determine the Tmax of enlicitide decanoate in Panel A, B, C and D participants. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis to report Tmax. Per protocol, mean Tmax was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 120, 168, and 240 hours postdose
Population: All participants of Panel A, B, C and D who received at least a dose of study treatment and had data available for Tmax.
Measure: Median (Full Range); unit: hours
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8
hours | 16 [1 to 24.25] | 2.75 [0.5 to 24] | 18.01 [0.50 to 48] | 1.00 [0.50 to 24] | 1.0 [0.5 to 12.03]

5. Primary Outcome: Apparent Terminal Half-life (t1/2) of Enlicitide Decanoate
Description: Half-life (t1/2) was defined as the time required for plasma drug concentration of enclitide decanoate to decrease by 50% from peak. Blood for plasma samples was collected at pre-specified time points to determine the t1/2 of enlicitide decanoate in Panel A, B, C and D participants. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis to report t1/2. Per protocol, mean t1/2 was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 120, 168, and 240 hours postdose
Population: All participants of Panel A, B, C, and D who received at least a dose of study treatment and had data available for the t1/2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 8
hours | 81.5 (70.4) | 56.4 (32.7) | 53.6 (36.9) | 75.6 (62.9) | 46 (60.8)

6. Primary Outcome: Apparent Clearance (CL/F) of Enlicitide Decanoate
Description: CL/F was the apparent total clearance of enlicitide decanoate in plasma over time. Blood for plasma samples was collected at pre-specified timepoints to determine the CL/F of enlicitide decanoate for Panel A, B, C, and D participants. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis to report CL/F. Per protocol, mean CL/F was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 120, 168, and 240 hours postdose
Population: All participants of Panel A, B, C, and D who received at least a dose of study treatment and had data available for the CL/F.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hr
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 8
Liter/hr | 17.6 [12 to 25.9] | 23.3 [15.9 to 34] | 15.2 [9.58 to 24] | 22.6 [16 to 31.9] | 26.5 [17.2 to 40.8]
Statistical Analysis 1: Comparison: Panel A: Moderate Renal Impairment (RI) vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.67, 90% CI 2-sided [0.43 to 1.02] — GMR and 90% CI were calculated using a linear fixed effects model performed on natural log-transformed values. GMR: Panel A-Moderate Renal Impairment (RI)/Panel D-Healthy controls
Statistical Analysis 2: Comparison: Panel B: Severe RI vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.88, 90% CI 2-sided [0.58 to 1.35] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geomtric Mean ratio = 0.57, 90% CI 2-sided [0.36 to 0.91] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geomtric Mean Ratio = 0.86, 90% CI 2-sided [0.57 to 1.29] — [estimate comment as in outcome 1, analysis 4]

7. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Enlicitide Decanoate
Description: Vz/F was the apparent volume of distribution of enlicitide decanoate between the plasma and the rest of the body, after dose, assessed as the total volume of enlicitide decanoate that would need to be uniformly distributed to achieve the desired plasma drug concentration. Blood for plasma samples was collected at pre-specified time points to determine the Vz/F of Enlicitide Decanoate in Panel A, B, C, and D participants. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis to report Vz/F. Per protocol, mean Vz/F was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 120, 168, and 240 hours postdose
Population: All participants of Panel A, B, C, and D who received at least a dose of study treatment and had data available for the Vz/F.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 8
Liter | 2070 [1370 to 3120] | 1890 [1300 to 2760] | 1170 [845 to 1620] | 2470 [1680 to 3620] | 1760 [1400 to 2210]
Statistical Analysis 1: Comparison: Panel A: Moderate Renal Impairment (RI) vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 1.18, 90% CI 2-sided [0.83 to 1.67] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Panel B: Severe RI vs Panel D: Healthy Controls; Test type: Other; Geometric Mean ratio = 1.08, 90% CI 2-sided [0.78 to 1.50] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.66, 90% CI 2-sided [0.50 to 0.89] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 1.40, 90% CI 2-sided [1.00 to 1.97] — GMR and 90% CI for AUC0-inf were calculated using a linear fixed effects model performed on natural log-transformed values. GMR: Panel C-ESRD Enlicitide Decanoate Post-Hemodialysis/ Panel D-Healthy Controls

8. Secondary Outcome: Panel C: Dialysate Clearance (CLd) of Enlicitide Decanoate
Description: CLd was the measure of the amount of enlicitide decanoate cleared from plasma via dialysis. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis. Urine samples were to be collected for Panel C participants to determine mean CLd.
Time Frame: Predose and 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, and 48 hours postdose
Population: Per protocol all participants of Panel C who received at least a dose of study treatment and had data available were to be analyzed. However, no urine samples could be collected on Panel C participants, thus no data were reported.
Arm/Group | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Panel C: Dialysate Concentration (Cd) of Enlicitide Decanoate
Description: Cd was the measure of the concentration of enlicitide decanoate in dialysate. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis. Urine samples were to be collected for Panel C participants to determine mean Cd.
Time Frame: Predose and 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, and 48 hours postdose
Population: as for outcome 8
Arm/Group | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-hemodialysis
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Panel C: Amount of Enlicitide Decanoate Excreted (AEd) in Dialysate
Description: AEd was the measure of the amount of enlicitide decanoate excreted in the dialysate. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis. Urine samples were to be collected for Panel C participants to determine mean AEd.
Time Frame: Predose and 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, and 48 hours postdose
Population: as for outcome 8
Arm/Group | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-hemodialysis
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Panel C: Percentage of Dose (%Dose) of Enlicitide Decanoate Excreted in Dialysate
Description: %Dose was the percentage of the dose of enlicitide decanoate excreted in the dialysate. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis. Urine samples were to be collected for Panel C participants to determine %Dose.
Time Frame: Predose and 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, and 48 hours postdose
Population: as for outcome 8
Groups:
- Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis: Participants received Enlicitide Decanoate 20 mg tablet single dose orally on Day 1.
- Panel C: ESRD - Enlicitide Decanoate Post-hemodialysis: Participants received Enlicitide Decanoate 20 mg tablet single dose orally on Day 16.
Arm/Group | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-hemodialysis
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Amount of Enlicitide Decanoate Excreted in Urine From 0 to 24 Hours (AE0-24) After Administration of Enlicitide Decanoate
Description: AE0-24 was the measure of the amount of enlicitide decanoate excreted at 0 to 24 hours. Urine samples were to be collected to determine the AE0-24 after administration of enlicitide decanoate for Panels A, B, C, and D. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis to report AE0-24. Per protocol, mean AE0-24 was reported.
Time Frame: Predose and 0, 0.5, 1, 1.5, 2, 4, 8, 12, and 24 hours postdose
Population: All participants from Panel A, B, C, and D who received a dose of study treatment and had data available for AE0-24 were to be analyzed. No urine samples were collected on Panel C participants; therefore, no data were reported for this group.
Measure: Geometric Mean (95% Confidence Interval); unit: mg
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 8 | 8 | 0 | 0 | 8
mg | 0.0213 [0.00846 to 0.0538] | 0.00592 [0.00211 to 0.0166] |  |  | 0.0662 [0.0371 to 0.118]
Statistical Analysis 1: Comparison: Panel A: Moderate Renal Impairment (RI) vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.32, 90% CI 2-sided [0.14 to 0.74] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Panel B: Severe RI vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.09, 90% CI 2-sided [0.04 to 0.22] — [estimate comment as in outcome 1, analysis 2]

13. Secondary Outcome: Percentage of Unchanged Enlicitide Decanoate Excreted in Urine (Fe)
Description: Fe was the measure of the percentage of unchanged enlicitide decanoate excreted in the urine. The percentage of enlicitide decanoate that was excreted unchanged in urine over the 24-hr collection interval (Fe) was calculated as 100 times the ratio of Ae0-24 and dose. Urine samples were to be collected to determine the Fe after administration of enlicitide decanoate for Panels A, B, C, and D. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis to report Fe.
Time Frame: Predose and 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, and 48 hours postdose
Population: All participants from Panel A, B, C, and D who received a dose of study treatment and had data available for Fe were to be analyzed. No urine samples were collected on Panel C participants; therefore, no data were reported for this group.
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of Enlicitide Decanoate
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 8 | 8 | 0 | 0 | 8
Percentage of Enlicitide Decanoate | 0.107 [0.0423 to 0.269] | 0.0296 [0.0105 to 0.0831] |  |  | 0.331 [0.185 to 0.591]
Statistical Analysis 1: Comparison: Panel A: Moderate Renal Impairment (RI) vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.32, 90% CI 2-sided [0.14 to 0.74] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Panel B: Severe RI vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.09, 90% CI 2-sided [0.04 to 0.22] — [estimate comment as in outcome 1, analysis 2]

14. Secondary Outcome: Renal Clearance (CLr) of Enlicitide Decanoate
Description: CLr was the measure of how quickly enlicitide decanoate was removed from the plasma by the kidney and excreted in urine. Urine samples were to be collected to determine the CLr after administration of enlicitide decanoate for Panels A, B, C, and D. Per protocol, Panel C ESRD on HD arm was separated into two arms: Panel C enlicitide decanoate pre-hemodialysis and Panel C enlicitide decanoate post-hemodialysis to report CLr. Per protocol, mean CLr was reported.
Time Frame: Predose and 0, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, and 48 hours postdose
Population: All participants from Panel A, B, C, and D who received a dose of study treatment and had data available for CLr were to be analyzed. No urine samples were collected on Panel C participants; therefore, no data were reported for this group.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hr
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: ESRD - Enlicitide Decanoate Pre-Hemodialysis | Panel C: ESRD - Enlicitide Decanoate Post-Hemodialysis | Panel D: Healthy Controls
Number analyzed (Participants) | 8 | 8 | 0 | 0 | 8
Liter/hr | 0.0716 [0.0349 to 0.147] | 0.0347 [0.0114 to 0.106] |  |  | 0.243 [0.161 to 0.366]
Statistical Analysis 1: Comparison: Panel A: Moderate Renal Impairment (RI) vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.29, 90% CI 2-sided [0.16 to 0.55] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Panel B: Severe RI vs Panel D: Healthy Controls; Test type: Other; Geometric Mean Ratio = 0.14, 90% CI 2-sided [0.06 to 0.36] — [estimate comment as in outcome 1, analysis 2]

15. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE were reported.
Time Frame: Up to approximately 30 days
Population: All allocated participants who received a dose of study treatment. Per protocol, AEs were not collected separately for Panel C ESRD - Enlicitide Decanoate pre-hemodialysis and Panel C ESRD Enlicitide Decanoate post-hemodialysis arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: End-Stage Renal Disease (ESRD) on Hemodialysis (HD) | Panel D: Healthy Controls
Number analyzed (Participants) | 8 | 8 | 9 | 8
Participants | 2 | 2 | 1 | 0

16. Secondary Outcome: Panels A, B, and D: Number of Participants Who Discontinued From the Study Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of Panel A, B, and D participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to approximately 30 days
Population: All allocated participants in Panels A, B and D who received a dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel D: Healthy Controls
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

17. Secondary Outcome: Panel C: Number of Participants Who Discontinued From the Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of Panel C participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to approximately 30 days
Population: All allocated participants in Panels C who received a dose of study treatment. Per protocol, AEs were not collected separately for Panel C ESRD - Enlicitide Decanoate pre-hemodialysis and Panel C ESRD Enlicitide Decanoate post-hemodialysis arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel C: End-Stage Renal Disease (ESRD) on Hemodialysis (HD)
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 30 days
Description: All-Cause Mortality reported for all allocated participants. Serious and non-serious adverse events (AEs) were reported on all allocated participants who received a dose of study treatment. Per protocol, All-cause mortality, serious and non-serious AEs were not collected separately for Panel C ESRD - Enlicitide Decanoate pre-hemodialysis and Panel C ESRD Enlicitide Decanoate post-hemodialysis arms.
Arm/Group | Panel A: Moderate Renal Impairment (RI) | Panel B: Severe RI | Panel C: End-Stage Renal Disease (ESRD) on Hemodialysis (HD) | Panel D: Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/9 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 2/8 | 0/9 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: Moderate Renal Impairment (RI) (N=8) | Panel B: Severe RI (N=8) | Panel C: End-Stage Renal Disease (ESRD) on Hemodialysis (HD) (N=9) | Panel D: Healthy Controls (N=8)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: Moderate Renal Impairment (RI) (N=8) | Panel B: Severe RI (N=8) | Panel C: End-Stage Renal Disease (ESRD) on Hemodialysis (HD) (N=9) | Panel D: Healthy Controls (N=8)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all manuscripts or abstracts before submission. Any information identified by the sponsor as confidential must be deleted prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT05934292/Prot_SAP_000.pdf